CLINICAL TRIAL: NCT04268732
Title: Causes of Acute Undifferentiated Fever and the Utility of Biomarkers in Differentiating Bacterial From Viral Infection Among Acute Febrile Patients in Northwest Ethiopia
Brief Title: Acute Undifferentiated Fever in Ethiopia
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Gondar (Other)
Responsible Party: Sponsor
Other Study IDs: 1284/19
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Acute Febrile Illness
Keywords: biomarkers; bacterial infection; viral infection; malarial infection
MeSH Terms: conditions — Bacterial Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood serum blood culture bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study on acute undifferentiated fever and the utility of biomarkers in differentiating bacterial from viral infection among acute febrile patients in Gondar, northwest Ethiopia.

DETAILED DESCRIPTION:
General objective:

To assess the causes of acute undifferentiated febrile illness and evaluation of biomarkers for differentiation of bacterial and viral infections among outpatients at University of Gondar (UOG) Hospital, Northwest Ethiopia

Specific objectives

1. To determine the number of malaria cases, bacterial infections (by blood culture and polymearase chain reaction (PCR) for Rickettsia and Borrelia), and arboviral infections (DENV, YFV, CHIKV) among all acute febrile patients
2. To evaluate the diagnostic performance different assays (RDT, RT-(reverse transcriptase)PCR, ELISA) for the diagnosis of DENV
3. To evaluate the qualitative detection of C-reactive protein (CRP) and Myxovirus resistance protein (MxA) (by FebriDx RDT) and quantitative CRP detection for differentiating bacterial and viral infections

Study design, population, materials and methods: a cross-sectional cohort study on febrile patients presenting with acute fever at the emergency ward of the UOG hospital from June to August 2019. Clinical and epidemiological data will be recorded in a pseudo-anonymized and collected using an electronic data collection tool (KoBoToolbox). Blood will be collected for RDT testing, blood culture, PCR and serum for ELISA and RT-PCR.

Sample size: 200 acute febrile patients

Expected results and relevance: Evaluation of the causes of acute febrile illness and the role of biomarkers in differentiating viral and bacterial infections will increase the awareness of circulating pathogens and improve patient management. This evidence will contribute to a more rational use of laboratory diagnostic tests, antibiotics and antimalarial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute fever (an axillary temperature of ≥37.5°C; symptom duration ≤7 days)
* ≥ 15 years old
* signed informed consent

Exclusion Criteria:

* pregnant woman & children (<15 y)
* febrile patient suspected of urinary tract infection or acute respiratory tract infection
* Individuals who had taken antimicrobial and antimalarial drug in the last 2 weeks
* Patients with acute injury or trauma or for which participation in the study implies an unacceptable health risk as determined by the physicians

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients ≥ 15 years old with acute undifferentiated fever and seeking health services within 7 days after fever onset at the emergency ward of the university of Gondar hospital (Ethiopia) during the study period.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The differentiation of bacterial infections and viral infections among acute febrile patients with biomarkers | within 7 days after onset of fever
  CRP (bacterial biomarker) and MxA (viral biomarker) will be evaluated for differentiating confirmed bacterial and viral infections.

SECONDARY OUTCOMES:
The number of malaria cases, bacterial infections, viral infections and unknown etiologies among acute febrile patients in Gondar | within 7 days after onset of fever
  Different diagnostic tools will be used for analysis of acute febrile patient samples to confirm malaria (by RDT), bacterial infection (by blood culture and PCR for Rickettsia and Borrelia) and for viral infections (by RT-PCR for DENV, CHIKV, YFV). Samples negative for all these tests are defined as unknown etiology.
The comparison of different assays for diagnosis of DENV | within 7 days after onset of fever
  Different diagnostic tests will be evaluated for the detection of acute DENV infection (NS1 RDT, RT-PCR, ELISA IgM) and past DENV infection (ELISA IgG) among acute febrile patients.
The comparison of the qualitative and qualitative detection of CRP for differentiating bacterial and viral infections | within 7 days after onset of fever
  Qualitative CRP levels will be measured by FebriDx test and quantitative CRP levels will be measured by QuikReadGo. The detection of > 20mg/L CRP will be used to evaluate the confirmed bacterial infections and to compare with antibiotic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Johan van Griensven, PhD, MD, Study Director — Institute of Tropical Medicine
Locations (2):
- Institute of Tropical Medicine, Antwerp, Belgium
- University of Gondar, Gonder, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhargava A, Ralph R, Chatterjee B, Bottieau E. Assessment and initial management of acute undifferentiated fever in tropical and subtropical regions. BMJ. 2018 Nov 29;363:k4766. doi: 10.1136/bmj.k4766. No abstract available. PMID 30498133
- [Background] Mohammed Yusuf A, Abdurashid Ibrahim N. Knowledge, attitude and practice towards dengue fever prevention and associated factors among public health sector health-care professionals: in Dire Dawa, eastern Ethiopia. Risk Manag Healthc Policy. 2019 Jun 7;12:91-104. doi: 10.2147/RMHP.S195214. eCollection 2019. PMID 31239796
- [Background] Ferede G, Tiruneh M, Abate E, Wondimeneh Y, Damtie D, Gadisa E, Howe R, Aseffa A, Tessema B. A serologic study of dengue in northwest Ethiopia: Suggesting preventive and control measures. PLoS Negl Trop Dis. 2018 May 31;12(5):e0006430. doi: 10.1371/journal.pntd.0006430. eCollection 2018 May. PMID 29852020
- [Background] Lilay A, Asamene N, Bekele A, Mengesha M, Wendabeku M, Tareke I, Girmay A, Wuletaw Y, Adossa A, Ba Y, Sall A, Jima D, Mengesha D. Reemergence of yellow fever in Ethiopia after 50 years, 2013: epidemiological and entomological investigations. BMC Infect Dis. 2017 May 15;17(1):343. doi: 10.1186/s12879-017-2435-4. PMID 28506254
- [Background] Animut A, Mekonnen Y, Shimelis D, Ephraim E. Febrile illnesses of different etiology among outpatients in four health centers in Northwestern Ethiopia. Jpn J Infect Dis. 2009 Mar;62(2):107-10. PMID 19305049
- [Background] Kapasi AJ, Dittrich S, Gonzalez IJ, Rodwell TC. Host Biomarkers for Distinguishing Bacterial from Non-Bacterial Causes of Acute Febrile Illness: A Comprehensive Review. PLoS One. 2016 Aug 3;11(8):e0160278. doi: 10.1371/journal.pone.0160278. eCollection 2016. PMID 27486746
- [Background] Self WH, Rosen J, Sharp SC, Filbin MR, Hou PC, Parekh AD, Kurz MC, Shapiro NI. Diagnostic Accuracy of FebriDx: A Rapid Test to Detect Immune Responses to Viral and Bacterial Upper Respiratory Infections. J Clin Med. 2017 Oct 7;6(10):94. doi: 10.3390/jcm6100094. PMID 28991170